CLINICAL TRIAL: NCT01349608
Title: Physical Activity Coaching in COPD
Brief Title: Physical Activity Coaching in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, Consultant Pulmonary and Critical Care Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-000356
Record Dates: First submitted 2011-05-02; First posted 2011-05-06 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Physical Activity; Health Behavior
Keywords: Chronic Obstructive Pulmonary Disease; Motivational Interviewing; Health Coaching; Physical Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health coaching (Experimental)
  Interventions: Behavioral: Telephonic health coaching

INTERVENTIONS:
Behavioral: Telephonic health coaching — Participants will be given a pedometer and activity log to use daily to track their physical activity accomplishments. Weekly, they will participate in a health coaching telephone session to discuss physical activity and set goals. The health coach is knowledgable in COPD care and will utilize a motivational interviewing approach to support the self-efficacy of the participants to be more active.

SUMMARY:
This study is designed to explore a new approach to help people with chronic obstructive pulmonary disease (COPD) become more physically active. Through weekly telephone sessions with a health coach utilizing motivational interviewing, participants will be empowered to set goals for increased physical activity (emphasis on walking). The objective of the study is to determine if telephone-based health coaching is a reasonable and effective way to increase physical activity, as measured by a gold-standard activity monitor, in people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 40 years and older
* Current or former cigarette smoker of at least 10 pack-years
* Diagnosis of COPD stage II to IV COPD as documented by pulmonary function testing (FEV1 <80% predicted, FEV1/FVC ration <0.71) within the past 24 months
* Able to ambulate independently or with a walking aid (wheeled or standard walker or cane)

Exclusion Criteria:

* Unable to walk without assistance of another person
* patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency), are planning to move out of the state, are not able to be contacted by telephone
* patients with an inability to provide good data or follow commands (patients who are disoriented or have a severe neurologic/psychiatric condition)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of telephone-based health coaching in COPD. | 3 Months
  Determine the effectiveness of a telephone-based health coaching intervention on daily physical activity level, as measured by a gold-standard activity monitor and daily pedometer record, acceptability of intervention through qualitative interviews with participants, and health-related quality of life as measured by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States